CLINICAL TRIAL: NCT01756690
Title: Endogenous Heparinoid Interference With Coagulation on Thromboelastogram as a Predictive Biomarker for Transfusion Related Acute Lung Injury (TRALI)
Brief Title: Predicting Lung Injury From Transfusion in Patients With Liver Disease
Status: Terminated | Type: Observational
Why Stopped: Recruitment
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0238
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Transfusion-related Acute Lung Injury; Chronic Liver Disease; Gastrointestinal Bleeding
Keywords: respiratory distress syndrome, adult; blood component transfusion; gastrointestinal hemorrhage; blood coagulation
MeSH Terms: conditions — Transfusion-Related Acute Lung Injury; Gastrointestinal Hemorrhage; Respiratory Distress Syndrome; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A certain molecule floating in the blood may represent a risk of lung injury after a transfusion. We are determining whether detection of this molecule on a simple blood clotting test will predict the development of lung injury due to transfusion in bleeding patients with chronic liver disease.

ELIGIBILITY:
Inclusion criteria: Subjects will be eligible to participate in the study if they meet all of the following criteria:

1. Admit to an ICU due to gastrointestinal bleeding AND an INR > 1.5
2. Patient has chronic liver disease defined as 1 or more of the three following diagnostic criteria:

   1. Previous diagnosis of chronic liver disease OR Imaging or biopsy diagnosis of cirrhosis
   2. Signs of portal hypertension (ascites, varices, hypersplenism)
   3. Laboratory evidence of synthetic dysfunction (INR>1.5, Bilirubin> 2.0, Albumin< 2.5) AND ≥2 physical exam findings on admission associated with chronic liver disease (palmar erythema, spider angiomata, asterixis, caput medusa, gynecomastia)

Exclusion criteria: Subjects will be ineligible to participate in the study if they meet any of the following criteria

1. Patient under age 18 OR pregnant OR incarcerated
2. Patient meets criteria for acute respiratory distress syndrome (ARDS) (PaO2/FiO2<165)
3. Patient admitted to ICU for re-bleed on same hospital admission OR has already received >4 units of plasma.
4. History of inheritable or acquired clotting or bleeding disorder
5. Patient actively anticoagulated or has recently received (within 72h) vitamin K antagonists, direct thrombin inhibitors, heparins or Xa antagonists

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic Liver disease admitted to an intensive care unit with a gastrointestinal bleed and INR> 1.5 who may receive plasma transfusion therapy.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
TRALI (consensus definition- with exception of absence of other acute lung injury risk factors) | 0-54 hours post enrollment

SECONDARY OUTCOMES:
Change in ratio of partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) | 0-54 hours post enrollment
Bleeding complications | 0-5 days post-enrollmnet
  Baveno V criteria

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Denver, Anshutz medical campus, Aurora, Colorado
  - Denver Health and Hospital, Denver, Colorado